CLINICAL TRIAL: NCT01584518
Title: B-type Natriuretic Peptide (BNP) as a Surrogate Marker Guiding Post-operative Fluid Off-loading
Brief Title: B-type Natriuretic Peptide as a Surrogate Marker Guiding Post-operative Fluid Off-loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-16126
Record Dates: First submitted 2012-04-11; First posted 2012-04-25 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Fluid Over-load
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHF peptide (Active Comparator): Diuresis based on CHF-P
  Interventions: Drug: Furosemide
- Non CHF peptide (Active Comparator): Diuresis based on clinical judgement without data for CHF-P
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Based on clinical standard per clinician
  Other Names: Brand name: Lasix

SUMMARY:
The long-range goal of this proposal is to decrease morbidity and mortality related to pulmonary edema and congestive heart failure (CHF) in post-operative patients. The short-range goal is to determine a mechanistic endpoint when therapy for impending heart failure can be initiated and terminated based on B-type natriuretic peptide (BNP) levels. The investigators propose to utilize changing levels of BNP as a surrogate marker for CHF.

DETAILED DESCRIPTION:
Creighton University Medical Center is 334-bed Level I Trauma Center that hosts a wide variety of surgical and trauma patients. Many of these patients, including and especially those with pre-existing cardiac morbidities, develop symptoms of congestive heart failure (CHF) following trauma or surgical intervention because of a combination of physiological factors including third spacing followed by self-diuresis, and decreased contractility post injury. Normally, following the onset of CHF, surgeons begin treatment based on their clinical judgment of hemodynamic parameters and radiographic findings. CHF is known to increase morbidity, mortality, hospital length of stay and overall expenditure to the health care system and preventative measures and directed treatment modalities have potential to improve patient care and healthcare economics.

BNP, also known as beta-natriuretic protein or CHF peptide, is a cardiac neuro-hormone synthesized by the cardiac myocytes. It is released as a preproBNP peptide of 134 amino acids and is cleaved into proBNP (108 amino acids) and a signal peptide of 26 amino acids. ProBNP is subsequently cleaved into BNP (32 amino acids) and the inactive N-terminal proBNP peptide (NBNP; 76 amino acids). The effects of BNP are vasodilation, natriuresis and diuresis1.

Left ventricular end-diastolic wall stress (EDWS) measurement and ejection fraction are well established surrogates to predict the onset of CHF but require the invasive procedure of cardiac catheterization.

The mainstay of the treatment of CHF is diuretic drugs to try to remove excess fluid from the patient. In this project we plan to identify patients at risk for CHF and divide them into two groups. In one group BNP will be used to guide diuretic dosage and in the other conventional clinical parameters will be used.

ELIGIBILITY:
Inclusion Criteria:

* General Surgery patients with history of coronary artery disease, congestive heart failure, pulmonary hypertension
* Cardiac surgery patients undergoing CABG (coronary artery bypass grafting) and valve replacements

Exclusion Criteria:

1. Recent myocardial infarction (within 3 months).
2. ASA class 4 and more.
3. Emergency surgeries.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjan J Talukdar, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHF Peptide | Non CHF Peptide
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF Peptide | Non CHF Peptide | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (10) | 70 (9) | 70 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: The subjects will be evaluated preoperatively and followed post-operatively until discharge from the hospital. Length of stay
Time Frame: From date of admission until date of discharge, assessed up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CHF Peptide | Non CHF Peptide
Number analyzed (Participants) | 25 | 25
days | 4 (3) | 6 (5)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | CHF Peptide | Non CHF Peptide
Serious Adverse Events (participants affected / at risk) | 0/25 | 4/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF Peptide (N=25) | Non CHF Peptide (N=25)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Death (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes